CLINICAL TRIAL: NCT03395093
Title: Bispectral Index Monitoring of Sedation Depth During Flexible Bronchoscopy: With or Without Fentanyl .
Brief Title: BIS of Sedation Depth During Flexible Bronchoscopy.
Acronym: BIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YL20160713-021
Record Dates: First submitted 2017-12-25; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Disease
Keywords: bronchoscopy; conscious sedation; fentanyl; Bispectral Index
MeSH Terms: conditions — Lung Diseases | interventions — Fentanyl; Midazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FB with fentanyl (Experimental): In the Bispectral Index monitoring,our study will use midazolam, propofol and fentanyl in the conscious sedation of FB
  Interventions: Drug: Fentanyl; Drug: Midazolam; Drug: Propofol; Device: Bispectral Index monitoring
- FB without fentanyl (Active Comparator): In the Bispectral Index monitoring, our study will use midazolam, propofol in the conscious sedation of FB
  Interventions: Drug: Midazolam; Drug: Propofol; Device: Bispectral Index monitoring

INTERVENTIONS:
Drug: Fentanyl — Five minutes before the patients is done the flexible bronchoscopy, fentanyl will be intravenous injected.
  Other Names: fentanest; fantail; sublimaze
  Arms: FB with fentanyl
Drug: Midazolam — Five minutes before the patients is done the flexible bronchoscopy, midazolam will be intravenous injected.
  Other Names: Ro-21-3981
Drug: Propofol — Propofol will be intravenous injected as soon as the flexible bronchoscopy begins.
  Other Names: diprivan; disoprofol
Device: Bispectral Index monitoring — Bispectral Index monitoring will be used in the process of the flexible bronchoscopy.

SUMMARY:
Fentanyl is analgesia medication. There has not pain nerve in the lung. Flexible bronchoscopy(FB) is used in the respiratory medicine. So people will not feel pain in the process of FB. The purpose of the study is to know if Fentanyl is useful in the conscious sedation of FB.

DETAILED DESCRIPTION:
Fentanyl is opioid receptor agonists. It is a fast-acting, short duration and potent analgesics.

Flexible bronchoscopy (FB) is mostly used in the diagnosis and therapy in the respiratory disease. As we know, there has not pain nerve in the lung. People will not feel pain when they are in FB.

If fentanyl will be effective in FB? Our study will observe the effect of conscious sedation in FB with fentanyl or without fentanyl.

ELIGIBILITY:
Inclusion Criteria:

Cough reflex is good agree to do bronchoscopy agree to take part in the study no the contraindication of bronchoscopy

Exclusion Criteria:

Forced expiratory volume in one second<1 L severe hemoptysis severe heart, liver,kidney failure psychiatric and nervous disorders allergic to the anesthetic ( fentanyl, midazolam, or propofol)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
perioperative changes of blood pressure | every 5 minutes from the operation beginning to end
  For each patient,bispectral index monitoring after anesthesia. Bp will be measured.

SECONDARY OUTCOMES:
perioperative time | from the operation beginning to end
  For each patient, record the time bronchoscopy in and out
Adverse events | in the process of the operation
  For each patient, Adverse events (overall intraoperative cough,bleeding,low oxygen solution) will be record in the operation
Patient satisfaction rate | One day after the operation
  One day after the patient do the bronchoscopy, ask him/her about the satisfaction to the operation

CONTACTS AND LOCATIONS:
Overall Officials: wei gu, master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clark G, Licker M, Younossian AB, Soccal PM, Frey JG, Rochat T, Diaper J, Bridevaux PO, Tschopp JM. Titrated sedation with propofol or midazolam for flexible bronchoscopy: a randomised trial. Eur Respir J. 2009 Dec;34(6):1277-83. doi: 10.1183/09031936.00142108. Epub 2009 May 14. PMID 19443532
- [Result] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- See also: Titrated sedation with propofol or midazolam for flexible bronchoscopy: a randomised trial. — https://www.ncbi.nlm.nih.gov/pubmed/19443532
- See also: American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. — https://www.ncbi.nlm.nih.gov/pubmed/?term=American+College+of+Chest+Physicians++Consensus+Statement+on+the+Use+of+Topical++Anesthesia%2C+Analgesia%2C+and+Sedation+During+Flexible+Bronchoscopy+in+Adult+Patients